CLINICAL TRIAL: NCT07315958
Title: A Multinational, Multicenter, Observational, Prospective Cohort Study for Assessing the Prevalence of Airflow Limitation in Outpatients With History of Smoking Attending Cardiology Clinics
Acronym: ALSAC
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00124
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Respiratory (Chronic Obstructive Pulmonary Disease)
Keywords: chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a global health concern, associated with structural lung abnormalities causing persistent airflow limitation (AL) and often result from cigarette smoking. In Turkey, COPD was ranked the third among the mortality causes and the eighth among disability causes, with 9.1% to 19.1% prevalence rate. In the Middle East and North Africa (MENA) region, an increase of 30.6% in age-standardized point prevalence occurred between 1990 and 2019, with an estimated 10.7 million COPD cases. Similarly, in the sub-Saharan Africa region, the highest COPD prevalence rate of 24.8% was observed in South Africa. And in Kenya, East Africa, the pooled point estimate prevalence of COPD was 11.3%. The prevalence of COPD varies substantially between countries, but comparing numbers is challenging because they are recorded in different units and during different periods.

Patients with COPD are more likely to develop cardiovascular disease (CVD). For instance, COPD has been shown to increase the risk of acute myocardial infarction by 40% and stroke by 50%. Likewise, COPD patients with CVD have a considerably higher risk of COPD exacerbations than those without CVD. COPD and CVD have been linked to a worse prognosis primarily related to increased systemic inflammation; the presence of a concomitant disease with COPD leads to reduced quality of life, increased hospitalizations, and worse survival. For instance, every increase of 70 cL/s in forced expiratory volume in 1 second (FEV1) reduces mortality risk by 28%-35% from cardiovascular disease and 68%-72% from respiratory disease. Besides that, smoking has been shown to increase the risk of myocardial infarction (MI) and heart failure (HF) twofold, cigarette smoking toxins promote inflammation systemically, which may result in emphysema and atherosclerosis. Nevertheless, chronic inhalation of irritants, including biomass fuel smoke and air pollutants, produces an innate immune response and a later activation of adaptive immunity that might further amplify inflammation. Similarly, age-related elastin degradation may increase the risk of emphysema and arterial hypertension. On the contrary, physical activity is associated with improved lung function and a lower resting heart rate (RHR); consequently, COPD and CVD are more prevalent in sedentary populations. Observational studies suggest that decreasing the progression of COPD may assist in preventing cardiovascular morbidity and mortality, which is related to more severe respiratory symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 40 years or older.
2. Patients with a smoking history of 10 pack-years or more.
3. Patients willing and able to complete pulmonary function test, using a spirometer.
4. Patients who have provided written consent to participate in the study.
5. Patients attending cardiology clinics at the participating centers.
6. Patients willing and able to complete the CAAT questionnaire.

Exclusion Criteria:

A. Patients diagnosed with bronchial asthma. B. Patients who used a bronchodilator for an acute respiratory infection before performing spirometry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending cardiology clinics for any reason:
  1. Patients aged 40 years or older.
  2. Patients with a smoking history of 10 pack-years or more.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence (number and percentage) of outpatients attending cardiology clinics, with a history of smoking who exhibit concurrent AL consistent with COPD. | 1 Year
  Prevalence (number and percentage) of outpatients attending cardiology clinics, with a history of smoking who exhibit concurrent AL consistent with COPD.

SECONDARY OUTCOMES:
The proportion of patients with CVD who were previously diagnosed with COPD. | 1 Year
  The proportion of patients with CVD who were previously diagnosed with COPD.
The distribution of patients with AL consistent with COPD among AL severity GOLD grades 1-4. | 1 Year
  The distribution of patients with AL consistent with COPD among AL severity GOLD grades 1-4.
CAAT score of patients with AL consistent with COPD. | 1 Year
  CAAT score of patients with AL consistent with COPD.
The severity of COPD | 1 year
  The severity of COPD using GOLD ABE assessment scheme.